CLINICAL TRIAL: NCT00985140
Title: A Phase II Study of Total Skin Electron Beam Therapy (TSEBT) to Dose of 12 Gy in Stage IB-IIIA Mycosis Fungoides
Brief Title: Phase 2 Total Skin Electron Beam Therapy (TSEBT 12 Gy) in Stage IB-IIIA Mycosis Fungoides
Status: Terminated | Type: Observational
Why Stopped: Competing studies
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Richard T. Hoppe, Henry S. Kaplan-Harry Lebeson Professor of Cancer Biology, Stanford University
Other Study IDs: IRB-16402; SU-09082009-3760 (Other: Stanford University); LYMNHL0072 (Other: OnCore)
Record Dates: First submitted 2009-09-24; First posted 2009-09-28 (Estimated); Results first posted 2017-04-04 (Actual); Last update posted 2017-06-02 (Actual); Status verified 2017-05

CONDITIONS: Mycosis Fungoides; Lymphomas: Non-Hodgkin; Lymphomas: Non-Hodgkin Peripheral T-Cell; Lymphomas: Non-Hodgkin Cutaneous Lymphoma
MeSH Terms: conditions — Mycosis Fungoides

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 2 x 5mm punch biopsies taken at enrollment and during follow up.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 12 Gy TSEBT: Prospective assignment to receive 12 Gy total skin electron beam therapy (TSEBT) for mycosis fungoides
  Interventions: Radiation: Total Skin Electron Beam Therapy (TSEBT)

INTERVENTIONS:
Radiation: Total Skin Electron Beam Therapy (TSEBT) — The purpose of the study is to examine the efficacy and safety of total skin electron beam therapy to a dose of 12 Gray (TSEBT 12 Gray) in patients who have mycosis fungoides (MF) staged as IB to IIIB.

SUMMARY:
To examine the efficacy and safety of total skin electron beam therapy to a dose of 12 Gray (TSEBT 12 Gy) in patients who have mycosis fungoides (MF) staged as IB to IIIA.

DETAILED DESCRIPTION:
Total skin electron beam therapy will be administered in the Department of Radiation Oncology according to the Stanford six-field technique. Patients will receive a planned total skin dose of 12 Gy fractionated at 2 Gy/cycle (each cycle requiring 2 days of treatment) 4 days each week, for 3 weeks. Supplements will routinely be applied to the perineum and soles as well as any other "shadowed" sites involved by disease, such as the inframammary regions (1-2 Gy fractions to a total dose of 12 Gy). Discrete tumors may receive additional "boost" treatment not to exceed 12 Gy. During the course of TSEBT patients will be evaluated weekly in the Department of Radiation Oncology for determination of adverse events and toxicity grading according the NCI Common Toxicity Criteria (CTC) Version 3.0.

A baseline evaluation will occur on the first day of TSEBT at which time the following procedures will be performed: (This visit may be waived if TSEBT is initiated within one week of the screening visit AND there is no clinical evidence of disease progression). After the completion of TSEBT, patients will be followed every 4 weeks until 24 weeks , and then every 8 weeks for a total of 12 months or until there is disease progression, relapse, or the initiation of a new anti-cancer therapy. Patients who withdraw during the treatment period due to intolerance to radiotherapy will be followed weekly until toxicities have reverted to Grade ≤ 2 or has stabilized in the opinion of the Investigator, at which point a final visit will be scheduled. A final visit should be attempted for all patients who are lost to follow-up.

ELIGIBILITY:
Inclusion Criteria:1. Biopsy-confirmed mycosis fungoides in stage IB-IIIA

2. Patients must have failed or have been intolerant to at least one prior systemic or topical therapy which may include topical steroids

3. 18 years of age or older

4. Life expectancy greater than 6 months

5. Eastern Cooperative Oncology Group (ECOG) of <= 2

6. Adequate bone marrow function: WBC> 2000/uL; platelet count> 75,000/mm3; ANC> 1000

7. Required wash out period for prior therapies (Note: patients with progressive disease may be treated earlier than required washout period per Investigator's decision)

* Topical therapy: 2 weeks
* Systemic biologic, monoclonal antibody or chemotherapy: 4 weeks
* Radiotherapy (excluding TSEBT) or phototherapy: 4 weeks
* Other investigational therapy: 4 weeks

  8. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:1. Prior courses of TSEBT (Note: localized skin-directed radiotherapy is allowed if administered at least 4 weeks prior to initiation on study)

2. Underlying medical condition including unstable cardiac disease, or other serious illness that would impair the ability of patient to undergo treatment

3. Prior malignancy (active within 5 years of screening) except completely excised non-invasive basal cell or squamous cell carcinoma of the skin, or in situ squamous cell carcinoma of the cervix

4. Pregnant or lactating

5. Initiation or change in dosage of topical corticosteroids within 3 weeks of study treatment (Note: topical steroid use within 3 weeks is allowed provided the strength and use has been stable for at least 1 month; "prescription strength"topical corticosteroids cannot be started during the study)

6. Any other medical history, including laboratory results, deemed by the Investigator to be likely to interfere with patient participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with mycosis fungoides refractory to at lest one prior treatment.
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2009-06; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard T. Hoppe, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- Available data/document: Peer reviewed article with pooled results. — https://www.ncbi.nlm.nih.gov/pubmed/25476993 — This publication contains data from this study as well as two other clinical trials. Analysis was done on data pooled from the three trials.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients who may be eligible for the trial will be approached by the Investigator and offered participation in the trial. During a clinic visit, the Investigator or co-Investigator will explain the study to the potential subject verbally, and will allow the potential subject ample opportunity to ask questions.
Pre-assignment Details: Patients will undergo the following procedures during the screening period: Medical Hx, H&P, Severity Weighted Assessment Tool (mSWAT) assessment, simulation/set-up for TSEBT, CT if needed, pruritus, hair, and nail assessment, standardized photos (global, nails, head: top, front, sides, back), and two 5 mm punch biopsies from an active MF lesion.
Groups:
- 12 Gy TSEBT: Total skin electron beam therapy will be administered in the Department of Radiation Oncology according to the Stanford six-field technique. Patients will receive a planned total skin dose of 12 Gy fractionated at 2 Gy/cycle (each cycle requiring 2 days of treatment) 4 days each week, for 3 weeks. Discrete tumors may receive additional "boost" treatment not to exceed 12 Gy. .
Period: Overall Study
Arm/Group | 12 Gy TSEBT
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- 12 Gy TSEBT: Total skin electron beam therapy will be administered in the Department of Radiation Oncology according to the Stanford six-field technique. Patients will receive a planned total skin dose of 12 Gy fractionated at 2 Gy/cycle (each cycle requiring 2 days of treatment) 4 days each week, for 3 weeks. Discrete tumors may receive additional "boost" treatment not to exceed 12 Gy.
Arm/Group | 12 Gy TSEBT
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.4 (15.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 10
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Clinical Response Rate
Description: After the completion of TSEBT, patients will be followed every 4 weeks until 24 weeks ,and then every 8 weeks for a total of 12 months or until there is disease progression, relapse, or the initiation of a new anti-cancer therapy.
  The primary endpoint for the trial was the clinical response rate as defined by the modified severity weighted assessment tool (mSWAT) Partial response was defined as 50% improvement in the mSWAT. Complete response was complete disappearance of disease.
Time Frame: 1 year
Population: All patients who completed treatment.
Measure: Number; unit: participants
Arm/Group | 12 Gy TSEBT
Number analyzed (Participants) | 13
participants
  Partial Response | 11
  Stable disease | 2

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for 1 year.
Arm/Group | 12 Gy TSEBT
All-Cause Mortality (participants affected / at risk) | 0/13
Serious Adverse Events (participants affected / at risk) | 1/13
Other Adverse Events (participants affected / at risk) | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 12 Gy TSEBT (N=13)
Syncope (Nervous system disorders) | 1 (1) — Pt experienced grade 3 syncopal episode at home with no sequelae after the event
Dermatology/Skin Other (Skin and subcutaneous tissue disorders) | 1 (1) — Grade 3 skin reaction and numerous erythematous, denuded lesions on the right lateral leg and foot, and left arm.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 12 Gy TSEBT (N=13)
Erythema (Skin and subcutaneous tissue disorders) | 5 (5)
Fatigue (General disorders) | 7 (7)
Alopecia (Skin and subcutaneous tissue disorders) | 12 (12)
Dry Skin (Skin and subcutaneous tissue disorders) | 1 (1)
Nail Changes (Skin and subcutaneous tissue disorders) | 6 (6)
Skin Infection (Skin and subcutaneous tissue disorders) | 3 (3)
desquamation (Skin and subcutaneous tissue disorders) | 2 (2)
edema, nos (General disorders) | 1 (1)
Pain (extremity) (Gastrointestinal disorders) | 6 (6)
Skin and subcutaneous tissue disorders-other (Skin and subcutaneous tissue disorders) | 2 (2) — Blistering

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes